CLINICAL TRIAL: NCT01174121
Title: A Phase II Study Using Short-Term Cultured, Autologous Tumor-Infiltrating Lymphocytes Following a Lymphodepleting Regimen in Metastatic Cancers Plus the Administration of Pembrolizumab
Brief Title: Immunotherapy Using Tumor Infiltrating Lymphocytes for Patients With Metastatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100166; 10-C-0166
Record Dates: First submitted 2010-07-31; First posted 2010-08-03 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-08-08

CONDITIONS: Metastatic Colorectal Cancer; Metastatic Pancreatic Cancer; Metastatic Ovarian Cancer; Metastatic Breast Carcinoma; Metastatic Endocrine Tumors/ Neuroendocrine Tumors
Keywords: Digestive Tract Cancers; Breast Cancer; Endocrine Tumors; Ovarian/Endometrial Cancer; Genitourinary Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Endometrial Neoplasms; Urogenital Neoplasms | interventions — pembrolizumab; fludarabine; Cyclophosphamide; aldesleukin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 1/CD8+ Enriched TIL (CLOSED) (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + young CD8+ enriched TIL + high-dose aldesleukin (CLOSED)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Aldesleukin; Biological: Young TIL
- 2/Unselected TIL (CLOSED) (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + young unselected TIL + high-dose aldesleukin (CLOSED)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Aldesleukin; Biological: Young TIL
- 3/Unselected TIL + Pembro Prior to Cells (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + young unselected TIL + high-dose aldesleukin + pembrolizumab prior to cell administration and 3 additional doses every 3 weeks following cell infusion
  Interventions: Drug: Pembrolizumab (Keytruda); Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Aldesleukin; Biological: Young TIL
- 4/Unselected TIL + Pembro at POD (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + young unselected TIL + high-dose aldesleukin + pembrolizumab within 4 weeks of progressive disease for up to 8 doses every 3 weeks
  Interventions: Drug: Pembrolizumab (Keytruda); Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Aldesleukin; Biological: Young TIL
- 5/Unselected TIL + Pembro Prior to Cells (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + young unselected TIL + high-dose aldesleukin + pembrolizumab prior to cell administration and 3 additional doses every 3 weeks following cell infusion
  Interventions: Drug: Pembrolizumab (Keytruda); Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Aldesleukin; Biological: Young TIL

INTERVENTIONS:
Drug: Pembrolizumab (Keytruda) — Arm 3 or 5: Pembrolizumab 2mg/kg IV over approximately 30 minutes on Days -2, 21, 42, and 63 Arm 4: Pembrolizumab 2mg/kg IV over approximately 30 minutes (for patients who meet progressive disease per RECIST criteria and have resolved major toxicities after cell infusion or anytime during the post-treatment
  evaluation period; starting within 4 weeks of progression; may receive up to 8 doses every 3 weeks).
  Arms: 3/Unselected TIL + Pembro Prior to Cells; 4/Unselected TIL + Pembro at POD; 5/Unselected TIL + Pembro Prior to Cells
Drug: Fludarabine — Days -7 to -3: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days.
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with Mesna 15 mg/kg/day X2 days over 1 hr.
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg IV (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses.)
Biological: Young TIL — Day 0: Cells will be infused intravenously (IV) on the Patient Care Unit over 20-30 minutes (one to four days after the last dose of fludarabine).

SUMMARY:
Background:

The NCI Surgery Branch has developed an experimental therapy that involves taking white blood cells from patients' tumors, growing them in the laboratory in large numbers, and then giving the cells back to the patient. These cells are called Tumor Infiltrating Lymphocytes, or TIL and we have given this type of treatment to over 200 patients with melanoma. Researchers want to know if TIL shrink s tumors in people with digestive tract, urothelial, breast, or ovarian/endometrial cancers. In this study, we are selecting a specific subset of white blood cells from the tumor that we think are the most effective in fighting tumors and will use only these cells in making the tumor fighting cells.

Objective:

The purpose of this study is to see if these specifically selected tumor fighting cells can cause digestive tract, urothelial, breast, or ovarian/endometrial tumors to shrink and to see if this treatment is safe.

Eligibility:

- Adults age 18-72 with upper or lower gastrointestinal, hepatobiliary, genitourinary, breast, ovarian/endometrial cancer, or glioblastoma refractory to standard chemotherapy.

Design:

Work up stage: Patients will be seen as an outpatient at the NIH clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed.

Surgery: If the patients meet all of the requirements for the study they will undergo surgery to remove a tumor that can be used to grow the TIL product.

Leukapheresis: Patients may undergo leukapheresis to obtain additional white blood cells. (Leukapheresis is a common procedure, which removes only the white blood cells from the patient.)

Treatment: Once their cells have grown, the patients will be admitted to the hospital for the conditioning chemotherapy, the TIL cells and aldesleukin. They will stay in the hospital for about 4 weeks for the treatment.

Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking. Follow up visits will take up to 2 days.

...

DETAILED DESCRIPTION:
Background:

* Metastatic digestive tract cancers, in particular esophageal, gastric, pancreatic, and hepatobiliary carcinomas, are associated with poor survival beyond five years and poor response to existing therapies.
* Data from the National Cancer Institute Surgery Branch (NCI-SB) and from the literature support that metastatic cancers are potentially immunogenic and that tumor-infiltrating

lymphocytes (TIL) can be grown and expanded from these tumors.

* In metastatic melanoma, TIL can mediate the regression of bulky disease at any site when administered to an autologous patient with high-dose aldesleukin (IL-2) following a nonmyeloablative, lymphodepleting preparative regimen.
* The recent young-TIL approach, in which TIL are minimally cultured in vitro, not selected for tumor recognition, before rapid expansion and infusion to metastatic melanoma patients, has led to objective response rates comparable to previous trials relying on TIL screened for tumor recognition, with no added toxicities.
* In pre-clinical models, the administration of an anti-PD-1 antibody enhances the anti-tumor activity of transferred T-cells.
* We propose to investigate the feasibility, safety, and efficacy of TIL adoptive transfer therapy in combination with pembrolizumab, administered either prior to cell administration or at the time of progressive disease, for metastatic cancers.

Objectives:

-Primary objective:

--With Amendment BB, to determine the rate of tumor regression in patients with metastatic cancer who receive autologous, minimally cultured TIL in conjunction with a non-myeloablative, lymphodepleting preparative regimen, high-dose aldesleukin, and anti-PD-1.

Eligibility:

Patients must be/have:

* Age greater than or equal to 18 years and less than or equal to 72 years
* Metastatic upper or lower gastrointestinal, hepatobiliary, genitourinary, breast, ovarian/endometrial cancer, or endocrine tumors including neuroendocrine tumors refractory to standard chemotherapy

Patients may not have:

* Concurrent major medical illnesses
* Severe hepatic function impairment due to liver metastatic burden
* Unpalliated biliary or bowel occlusion, cholangitis, or digestive tract bleeding
* Any form of immunodeficiency
* Severe hypersensitivity to any of the agents used in this study

Design:

* Patients may undergo resection or biopsy to obtain tumor for generation of autologous TIL cultures and autologous cancer cell lines, and for frozen tissue archive. Lymph nodes, ascites,peritoneal implants, and normal tissue adjacent to metastatic deposit will also be obtained when possible for ongoing and future research as described in the NCI-SB cell harvest protocol 03-C-0277 (Cell Harvest and Preparation for Surgery Branch Adoptive Cell Therapy Protocols).
* With the approval of Amendment BB, patients will be enrolled on Arm 3 or Arm 4. All patients will receive a non-myeloablative, lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the infusion of autologous TIL and high-dose aldesleukin. Patients enrolled on Arm 3 will receive pembrolizumab prior to cell administration and three additional doses every three weeks following the cell infusion. Patients enrolled on Arm 4 will receive pembrolizumab within four weeks after meeting progressive disease by RECIST criteria, continuing for up to 8 doses every 3 weeks.
* Clinical and immunologic response will be evaluated about 6 weeks after cell infusion and periodically thereafter.
* Twenty-one patients will initially be enrolled in each group to assess toxicity and tumor responses. If two or more of the first 21 patients per groups shows a clinical response (partial response or complete response), accrual will continue to 41 patients, targeting a 20% goal for objective response.
* Up to 332 patients may be enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Measurable (per RECIST v1.0 criteria), metastatic cancer of one of the following types: upper or lower gastrointestinal, hepatobiliary, genitourinary, breast, ovarian/endometrial, or endocrine tumors including neuroendocrine tumors. Patients must have at least one lesion that is resectable for TIL generation with minimal morbidity, preferentially using minimal invasive laparoscopic or thoracoscopic surgery for removal of superficial tumor deposit.
* Confirmation of diagnosis of metastatic cancer by the NCI Laboratory of Pathology.
* Refractory to approved standard systemic therapy. Specifically:

  * Patients with metastatic colorectal cancer must have received oxaliplatin or irinotecan.
  * Patients with hepatocellular carcinoma must have received sorafenib (Nexavar(R)), since level 1 data support a survival benefit with this agent.
  * Patients with breast and ovarian cancer must be refractory to both first- and second-line treatments and must have received at least one second-line chemotherapy regimen.
* Patients with 3 or fewer brain metastases that are < 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for one month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
* Age greater than or equal to 18 years and less than or equal to 72 years.
* Clinical performance status of ECOG 0 or 1.
* Patients of both sexes must be willing to practice birth control from the time of enrollment on this study and 12 months after the last dose of combined chemotherapy for individuals of child-bearing potential (IOCBP) and for four months after treatment for individuals that can father children.
* IOCBP must have a negative pregnancy test be a pregnancy test prior to the start of treatment because of the potentially dangerous effects of the treatment on the fetus.

Serology

* Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive may have decreased immune-competence and thus may be less responsive to the experimental treatment and more susceptible to its toxicities.)
* Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then the patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.

Hematology

* ANC > 1000/mm^3 without the support of filgrastim
* WBC greater than or equal to 2500/mm^3
* Platelet count greater than or equal to 80,000/mm^3
* Hemoglobin > 8.0 g/dL. Subjects may be transfused to reach this cut-off.

Chemistry

* Serum ALT/AST less than or equal to 5.0 x ULN
* Serum creatinine less than or equal to 1.5 x ULN
* Total bilirubin less than or equal to 2.0 mg/dL, except in patients with Gilbert s Syndrome, who must have a total bilirubin < 3.0 mg/dL.
* Patients must have completed any prior systemic therapy at the time of enrollment.

Note: Patients may have undergone minor surgical procedures or limited field radiotherapy within the four weeks prior to enrollment, as long as related major organ toxicities have recovered to less than or equal to grade 1.

* Ability of subject to understand and the willingness to sign a written informed consent document.
* Willing to sign a durable power of attorney.
* Subjects must be co-enrolled on protocol 03-C-0277.

EXCLUSION CRITERIA:

* Participants who are pregnant or nursing because of the potentially dangerous effects of the treatment on the fetus or infant.
* Concurrent systemic steroid therapy.
* Active systemic infections requiring anti-infective treatment, coagulation disorders, or any other active or uncompensated major medical illnesses.
* Advanced primary with impeding occlusion, perforation or bleeding, dependent on transfusion.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and AIDS).
* History of major organ autoimmune disease.
* Grade 3 or 4 major organ irAEs clinically attributed to anti-PD-1/PD-L1 therapy.
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immunecompetence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
* History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, or aldesleukin.
* History of coronary revascularization or ischemic symptoms.
* For select patients with a clinical history prompting cardiac evaluation: last known LVEF less than or equal to 45%.
* Documented Child-Pugh score of B or C for hepatocellular carcinoma patients with known underlying liver dysfunction.
* For select patients with a clinical history prompting pulmonary evaluation: known FEV1 less than or equal to 50%.
* Patients who are receiving any other investigational agents.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2010-08-26 (Actual); Primary Completion 2028-12-27 (Estimated); Study Completion 2029-12-27 (Estimated)

PRIMARY OUTCOMES:
Response rate | 6 and 12 weeks after cell infusion, then every 3 months x3, then every 6 months x 2 years, then per PI discretion
  Percentage of patients who have a clinical response to treatment (objective tumor regression)

SECONDARY OUTCOMES:
Safety and efficacy of pembrolizumab in combination with TIL therapy | Every 6 weeks (week 6, 12, 18, 24) within 24 hours prior to next scheduled pembrolizumab dose
  Response rate and evaluation of treatment-related adverse events for patients who receive pembrolizumab
Frequency and severity of treatment-related adverse events | 30 days after end of treatment
  Aggregate of all adverse events, as well as their frequency and severity

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Chiba T, Ohtani H, Mizoi T, Naito Y, Sato E, Nagura H, Ohuchi A, Ohuchi K, Shiiba K, Kurokawa Y, Satomi S. Intraepithelial CD8+ T-cell-count becomes a prognostic factor after a longer follow-up period in human colorectal carcinoma: possible association with suppression of micrometastasis. Br J Cancer. 2004 Nov 1;91(9):1711-7. doi: 10.1038/sj.bjc.6602201. PMID 15494715
- [Background] Fong Y, Fortner J, Sun RL, Brennan MF, Blumgart LH. Clinical score for predicting recurrence after hepatic resection for metastatic colorectal cancer: analysis of 1001 consecutive cases. Ann Surg. 1999 Sep;230(3):309-18; discussion 318-21. doi: 10.1097/00000658-199909000-00004. PMID 10493478
- [Background] Tomlinson JS, Jarnagin WR, DeMatteo RP, Fong Y, Kornprat P, Gonen M, Kemeny N, Brennan MF, Blumgart LH, D'Angelica M. Actual 10-year survival after resection of colorectal liver metastases defines cure. J Clin Oncol. 2007 Oct 10;25(29):4575-80. doi: 10.1200/JCO.2007.11.0833. PMID 17925551
- [Derived] Lowery FJ, Goff SL, Gasmi B, Parkhurst MR, Ratnam NM, Halas HK, Shelton TE, Langhan MM, Bhasin A, Dinerman AJ, Dulemba V, Goldlust IS, Gustafson AM, Hakim AA, Hitscherich KJ, Kenney LM, Levy L, Rault-Wang JG, Bera A, Ray S, Seavey CD, Hoang CD, Hernandez JM, Gartner JJ, Sindiri S, Prickett TD, McIntyre LS, Krishna S, Robbins PF, Klemen ND, Kwong MLM, Yang JC, Rosenberg SA. Neoantigen-specific tumor-infiltrating lymphocytes in gastrointestinal cancers: a phase 2 trial. Nat Med. 2025 Jun;31(6):1994-2003. doi: 10.1038/s41591-025-03627-5. Epub 2025 Apr 1. PMID 40169866
- [Derived] Levin N, Kim SP, Marquardt CA, Vale NR, Yu Z, Sindiri S, Gartner JJ, Parkhurst M, Krishna S, Lowery FJ, Zacharakis N, Levy L, Prickett TD, Benzine T, Ray S, Masi RV, Gasmi B, Li Y, Islam R, Bera A, Goff SL, Robbins PF, Rosenberg SA. Neoantigen-specific stimulation of tumor-infiltrating lymphocytes enables effective TCR isolation and expansion while preserving stem-like memory phenotypes. J Immunother Cancer. 2024 May 30;12(5):e008645. doi: 10.1136/jitc-2023-008645. PMID 38816232
- [Derived] Zacharakis N, Huq LM, Seitter SJ, Kim SP, Gartner JJ, Sindiri S, Hill VK, Li YF, Paria BC, Ray S, Gasmi B, Lee CC, Prickett TD, Parkhurst MR, Robbins PF, Langhan MM, Shelton TE, Parikh AY, Levi ST, Hernandez JM, Hoang CD, Sherry RM, Yang JC, Feldman SA, Goff SL, Rosenberg SA. Breast Cancers Are Immunogenic: Immunologic Analyses and a Phase II Pilot Clinical Trial Using Mutation-Reactive Autologous Lymphocytes. J Clin Oncol. 2022 Jun 1;40(16):1741-1754. doi: 10.1200/JCO.21.02170. Epub 2022 Feb 1. PMID 35104158
- [Derived] Malekzadeh P, Pasetto A, Robbins PF, Parkhurst MR, Paria BC, Jia L, Gartner JJ, Hill V, Yu Z, Restifo NP, Sachs A, Tran E, Lo W, Somerville RP, Rosenberg SA, Deniger DC. Neoantigen screening identifies broad TP53 mutant immunogenicity in patients with epithelial cancers. J Clin Invest. 2019 Mar 1;129(3):1109-1114. doi: 10.1172/JCI123791. Epub 2019 Feb 4. No abstract available. PMID 30714987
- [Derived] Tran E, Turcotte S, Gros A, Robbins PF, Lu YC, Dudley ME, Wunderlich JR, Somerville RP, Hogan K, Hinrichs CS, Parkhurst MR, Yang JC, Rosenberg SA. Cancer immunotherapy based on mutation-specific CD4+ T cells in a patient with epithelial cancer. Science. 2014 May 9;344(6184):641-5. doi: 10.1126/science.1251102. PMID 24812403
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-C-0166.html